CLINICAL TRIAL: NCT02825953
Title: Does The Surfactant Administration by Aerosolization of Respiratory Distress Syndrome Effective in Spontaneously Breathing Premature Infants ?
Brief Title: Does The Surfactant Administration by Aerosolization Effective?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: nihat demir (Other)
Responsible Party: Sponsor-Investigator, nihat demir, Principal Investigator, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YYU-09
Record Dates: First submitted 2016-06-16; First posted 2016-07-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Respiratory Distress Syndrome; Surfactant Administration by Aerosolization
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Surface-Active Agents; poractant alfa; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nebulized surfactant (Active Comparator): For randomisatio, each infant will be randomly assigned to nasal continuous positive airway pressure (NCPAP) or non-invasive intermittent positive-pressure ventilation (NIPPV), and than premature babies with RDS breathing spontaneously will be administered surfactant by nebulizer.
  Interventions: Drug: surfactant; Device: nasal continuous positive airway pressure; Device: non-invasive intermittent positive-pressure ventilation; Device: Neopuff; Device: neonatal ventilator
- Endotracheal bolus application (Active Comparator): For randomisatio, each infant will be randomly assigned to nasal continuous positive airway pressure (NCPAP) or non-invasive intermittent positive-pressure ventilation (NIPPV). The investigators will administer surfactant via fundamental method.
  Interventions: Drug: surfactant; Device: nasal continuous positive airway pressure; Device: non-invasive intermittent positive-pressure ventilation; Device: Neopuff; Device: neonatal ventilator
- Minimally invasive surfactant therapy (Active Comparator): For randomisatio, each infant will be randomly assigned to nasal continuous positive airway pressure (NCPAP) or non-invasive intermittent positive-pressure ventilation (NIPPV). After randomisation, the investigators will administer surfactant via minimally invasive surfactant therapy (MIST) method which is recently very popular method
  Interventions: Drug: surfactant; Device: nasal continuous positive airway pressure; Device: non-invasive intermittent positive-pressure ventilation; Device: Neopuff; Device: neonatal ventilator

INTERVENTIONS:
Drug: surfactant — the investigators attempt to administer surfactant in a more gentle way, i.e. by nebulization, by minimally invasive surfactant therapy, and endotracheal bolus application of natural surfactant
  Other Names: Curosurf
Device: nasal continuous positive airway pressure — each infant will be randomly assigned to nasal continuous positive airway pressure (NCPAP) or non-invasive intermittent positive-pressure ventilation (NIPPV). The infants will be stabilised on NCPAP (Neopuff; Fisher and Paykel, Auckland, New Zealand) in the delivery room and during transport to the NICU. NCPAP or NIPPV will be started within 30 min of birth immediately after randomisation. Both NCPAP and NIPPV will be delivered by a neonatal ventilator (Engström Carestation; GE Healthcare, Madison, USA) via short, binasal Cannula (RAM Cannula; Neotech, Valencia, CA).
  Other Names: NCPAP
Device: non-invasive intermittent positive-pressure ventilation — each infant will be randomly assigned to nasal continuous positive airway pressure (NCPAP) or non-invasive intermittent positive-pressure ventilation (NIPPV). The infants will be stabilised on NCPAP (Neopuff; Fisher and Paykel, Auckland, New Zealand) in the delivery room and during transport to the NICU. NCPAP or NIPPV will be started within 30 min of birth immediately after randomisation. Both NCPAP and NIPPV will be delivered by a neonatal ventilator (Engström Carestation; GE Healthcare, Madison, USA) via short, binasal Cannula (RAM Cannula; Neotech, Valencia, CA).
  Other Names: NIPPV
Device: Neopuff — Fisher and Paykel, Auckland, New Zealand
Device: neonatal ventilator — GE Healthcare, Madison, USA
  Other Names: Engström Carestation

SUMMARY:
The present study was designed to evaluate, in premature babies with RDS breathing spontaneously, the efficacy of combined treatment with nasal continuous positive airway pressure (CPAP) and aerosolized surfactant. The first objective of investigators is to assess the safety of surfactant nebulization in this clinical situation, and to ﬁnd out whether treatment with aerosolized surfactant would reduce the need for mechanical ventilation. And other aim suggest that aerosolized dates compared with dates of INSURE (intubation-surfactant-extubation) and minimally invasive surfactant therapy (MIST) method.

DETAILED DESCRIPTION:
Does The Surfactant Administration by Aerosolization of Respiratory Distress Syndrome effective in Spontaneously Breathing Premature Infants ? Endotracheal bolus application of natural surfactant has been shown to be an effective treatment for idiopathic respiratory distress syndrome (RDS), especially in premature neonates with weeks of pregnancy > 27 week. However, patients are intubated nasotracheal or orotracheal for this form of treatment. This intubation carries potential risks of injuries to the dental lamina, the larynx, and the trachea, bronchopulmonary infections, and fluctuations in cerebral blood flow, intra- and periventricular haemorrhage (1). In addition, many babies with RDS who initially respond to surfactant therapy later develop chronic lung disease (CLD) (2). With this in mind, the investigators attempt to administer surfactant in a more gentle way, i.e. by nebulization. Administration by aerosol during spontaneous respiration is less traumatic and avoids intubation with the accompanying mechanical and infectious risks and pathophysiological effects.

The present study was designed to evaluate, in premature babies with RDS breathing spontaneously, the efficacy of combined treatment with nasal continuous positive airway pressure (CPAP) and aerosolized surfactant. The first objective of investigators is to assess the safety of surfactant nebulization in this clinical situation, and to ﬁnd out whether treatment with aerosolized surfactant would reduce the need for mechanical ventilation. And other aim suggest that aerosolized dates compared with dates of INSURE (intubation-surfactant-extubation) and minimally invasive surfactant therapy (MIST) method.

Seventy-five newborn babies from neonatal intensive care unit (NICU) of Yuzuncu Yil University Medical Scholl (Van, Turkey) will be randomized to treatment with nebulized surfactant (Curosurf®, Chiesi Pharmaceutics, Parma, Italy) or to two control groups receiving INSURE and MIST method. The study will be conducted with 75 infants, 25 in each group. Randomization will be central and performed using sealed envelopes kept at the neonatal ward of Yuzuncu Yil University Medical Centre Hospital. Informed consent was obtained from all parents before randomization. Inclusion criteria are corrected gestational age >26 week or <34 week, age 2-36 h, clinically and radiologically diagnosed progressive RDS, FiO2 needed to maintain SaO2 85-95%; >0.4, and no evident lung or cardiovascular malformation.

The surfactant aerosol will generate with a ultrasonic nebulizer (Aeroneb Pro; Aerogen, Inc., Sunnyvale, CA) and administer via the nasal continuous positive airway pressure (NCPAP) equipment into the Laryngeal Mask Airway (LMA). Surfactant will be diluted to 40 mg/ml with saline before nebulization. These modifications will be introduced to enhance the delivery of nebulized material to the lungs (3). In the control groups, the babies will be supported with the same type of NCPAP equipment, after given surfactant via endotracheal bolus application and MIST method. Parameters will be documented at three different times, namely before application of surfactant (200 mg/kg BW), and 2 h, 6 h after completion of nebulization or application of others.

The infants will be stabilised on NCPAP (Neopuff; Fisher and Paykel, Auckland, New Zealand) in the delivery room and during transport to the NICU. NCPAP or NIPPV will be started within 30 min of birth immediately after randomisation. Both NCPAP and NIPPV will be delivered by a neonatal ventilator (Engström Carestation; GE Healthcare, Madison, USA) via short, binasal Cannula (RAM Cannula; Neotech, Valencia, CA). NCPAP pressure will be set at 5-6 cm H2O, and NIPPV will be set in a non-synchronised mode at 20-30 bpm, with positive end-expiratory pressure of 5-6 cm H2O and peak inspiratory pressure of 15-20 cm H2O. FiO2 will be titrated at 0.21-0.50 to maintain an oxygen saturation level of 90%-95%, as measured via pulse oximeter. Under non-invasive ventilation, the surfactant will be administered as a rescue therapy if the infant required ≥0.40 FiO2 to maintain the target saturation level of 90%-95%.

Findings in chest radiograms before inclusion and head ultrasound images taken as soon as possible according to the clinical situation will be evaluated and graded according to criteria defined by Papile et al. (4) and Kero et al.(5) CLD will be defined as need for supplemental oxygen at 36 wk gestational age.

Statistical evaluation Data will be analyzed using the 20 Windows Version of Statistical Package for the Social Sciences (SPSS) Program (Chicago, IL, USA).

Data were compared using unpaired t-test and Chi-square test, and p-values below <0.05 were considered statistically significant.

Ethical approval The study was approved by the regional ethics committee at the Yuzuncu Yil University Institute, Van, Turkey.

The regional ethics committee No: 05.05.2015/09

ELIGIBILITY:
Inclusion Criteria:

* Corrected gestational age >26 week or <34 week,
* Age 2-36 h
* Clinically and radiologically diagnosed progressive RDS,
* FiO2 needed to maintain SaO2 85-95%; >0.4
* No evident lung or cardiovascular malformation.

Exclusion Criteria:

* Corrected gestational age <26 week or >34 week,
* Age >36 h
* Premature babies with RDS but no breathing spontaneously
* Evident lung or cardiovascular malformation.

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The first objective of investigators is to assess the safety of surfactant nebulization in this clinical situation, and to ﬁnd out whether treatment with aerosolized surfactant would reduce the need for mechanical ventilation. | within the ﬁrst 72 hour of life
  The infants will be stabilised on NCPAP (Neopuff; Fisher and Paykel, Auckland, New Zealand) in the delivery room and during transport to the NICU. NCPAP or NIPPV will be started within 30 min of birth immediately after randomisation. Both NCPAP and NIPPV will be delivered by a neonatal ventilator (Engström Carestation; GE Healthcare, Madison, USA) via short, binasal Cannula (RAM Cannula; Neotech, Valencia, CA). NCPAP pressure will be set at 5-6 cm H2O, and NIPPV will be set in a non-synchronised mode at 20-30 bpm, with positive end-expiratory pressure of 5-6 cm H2O and peak inspiratory pressure of 15-20 cm H2O. FiO2 will be titrated at 0.21-0.50 to maintain an oxygen saturation level of 90%-95%, as measured via pulse oximeter. Under non-invasive ventilation, the surfactant will be administered as a rescue therapy if the infant required ≥0.40 FiO2 to maintain the target saturation level of 90%-95%.

SECONDARY OUTCOMES:
Chronic Lung Disease (CLD) | up to 36 weeks of post gestational age
  Chronic Lung Disease (CLD) will be defined according to National Institutes of Health criteria.
Patent ductus arteriosus | In 5 days of life
  Echocardiography will be performed routinely for patent ductus arteriosus at a postnatal age of 48-96 h.
Intraventricular haemorrhage | Within 1 month of life
  We will assess for intraventricular haemorrhage higher than grade II using the Papile classification system
Necrotising enterocolitis | Within 3 months of life
  Necrotising enterocolitis with the modified Bell's classification system
Retinopathy of prematurity (ROP) | Up to 3 months of life
  Retinopathy of prematurity (ROP) requiring laser treatment based on the criteria of the American Academy of Pediatrics, American Academy of Ophthalmology and American Association for Pediatric Ophthalmology and Strabismus.

REFERENCES:
- [Result] Cowan F, Whitelaw A, Wertheim D, Silverman M. Cerebral blood flow velocity changes after rapid administration of surfactant. Arch Dis Child. 1991 Oct;66(10 Spec No):1105-9. doi: 10.1136/adc.66.10_spec_no.1105. PMID 1750756
- [Result] Mercier CE, Soll RF. Clinical trials of natural surfactant extract in respiratory distress syndrome. Clin Perinatol. 1993 Dec;20(4):711-35. PMID 8131364
- [Result] Berggren E, Liljedahl M, Winbladh B, Andreasson B, Curstedt T, Robertson B, Schollin J. Pilot study of nebulized surfactant therapy for neonatal respiratory distress syndrome. Acta Paediatr. 2000 Apr;89(4):460-4. doi: 10.1080/080352500750028195. PMID 10830460
- [Result] Papile LA, Burstein J, Burstein R, Koffler H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr. 1978 Apr;92(4):529-34. doi: 10.1016/s0022-3476(78)80282-0. PMID 305471
- [Result] Kero PO, Makinen EO. Comparison between clinical and radiological classification of infants with the respiratory distress syndrome (RDS). Eur J Pediatr. 1979 Apr 3;130(4):271-8. doi: 10.1007/BF00441363. PMID 436851